CLINICAL TRIAL: NCT01258868
Title: Epigenetically-Modified Autologous Tumor Cell Vaccines With ISCOMATRIX(TM) Adjuvant and Oral Celecoxib in Patients Undergoing Resection of Lung and Esophageal Cancers, Thymic Neoplasms, Thoracic Sarcomas, and Malignant Pleural Mesotheliomas
Brief Title: Tumor Cell Vaccines With ISCOMATRIX Adjuvant and Celecoxib in Patients Undergoing Resection of Lung and Esophageal Cancers and Malignant Pleural Mesotheliomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110041; 11-C-0041
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2016-08-17

CONDITIONS: Mesolthelioma; Esophageal Cancer; Lung Cancer; Thoracic Sarcomas; Thymoma
Keywords: Mesothelioma; Esophageal Cancer; Lung Cancer; Thoracic Malignancies; Tumor Cell Vaccine
MeSH Terms: conditions — Esophageal Neoplasms; Lung Neoplasms; Thymoma; Mesothelioma | interventions — Celecoxib; FANG vaccine

ARMS (1):
- 1 (Experimental): Celebrex+ tumor cell vaccine
  Interventions: Drug: Celebrex; Biological: Tumor cell vaccine

INTERVENTIONS:
Drug: Celebrex — 400 mg PO BID for 7 days prior to cell administration and then on days 1 through 28 of each vaccine cycle.
Biological: Tumor cell vaccine — A minimum of 1x10e7 and a maximum of 1x10e8 patient tumor cells that have been exposed to 1 mcM decitabine for 6 days, exposed to 100 Gy radiation and emulsified in 0.5 ml of the ISCOMATRIX adjuvant at a concentration of 180 ISCO units/mL administered IM every 4 weeks for 6 injections; if subject shows immune response, vaccine will be given every three months from months 9 - 24

SUMMARY:
Background:

- Recent research has shown that causing an immune response to tumor cells may help slow or stop the growth of tumors. One treatment that has come from this research involves collecting and modifying a cancer patient's tumor cells in the laboratory, then returning the cells to the patient as a vaccine to encourage the immune system to respond to them. Researchers are interested in testing tumor cell vaccines with an experimental drug called ISCOMATRIX , which can be added to a vaccine in order to elicit a stronger immune response in the body. ISCOMATRIX has not been approved for sale and use in any country and its use is still experimental, though it has been tested and used safely in other clinical studies. Researchers are also interested in determining whether the anti-inflammatory drug celecoxib will improve the body's immune reaction if given with the vaccine.

Objectives:

- To assess the safety and effectiveness of tumor cell vaccines given with ISCOMATRIX and celecoxib in the treatment of lung and esophagus cancers.

Eligibility:

* Individuals at least 18 years of age who have primary small cell or non-small cell lung cancer, esophageal cancer, or pleural mesothelioma that can be removed by surgery.
* Only individuals whose tumor cells are able to produce a tumor cell line for vaccine development will be eligible for treatment.

Design:

* Participants will be screened with a physical examination and medical history, and will have tumor tissue collected during their surgery to determine whether the tumor cells can be used to produce a vaccine.
* Participants will take celecoxib twice daily for 7 days before having the first tumor cell vaccination. Participants will also have leukapheresis to collect blood cells for testing before the first vaccination.
* Participants will receive one vaccine (which may be given in two shots) monthly for 6 months, and will continue to take celecoxib twice daily. One month after the 6th vaccine shot, participants will have another leukapheresis and skin test. If these tests show that a participant is responding to the vaccine, additional vaccines will be given every 3 months for up to 2 years.
* Participants will have a physical exam and lab tests before each vaccination, blood samples and imaging studies every 3 months, and a skin test every 6 months.
* Participants will have regular followup visits with imaging studies and blood samples for up to 5 years after the first vaccination, or until a new tumor develops.

DETAILED DESCRIPTION:
Background:

* Cancer-testis (CT) antigens have emerged as attractive targets for cancer immunotherapy. Whereas lung and esophageal cancers, thymic Neoplasms, primary thoracic sarcomas, as well as malignant pleural mesotheliomas express a variety of CT antigens, primary or vaccine-induced immune responses to these antigens appear uncommon in patients with these malignancies, possibly due to low-level, heterogeneous antigen expression, and inadequate vaccination strategies.
* Because numerous CT antigens can be induced in tumor cells by DNA demethylating agents and HDAC inhibitors, it is conceivable that vaccination of cancer patients with autologous tumor cells exposed to chromatin remodeling agents will enhance anti-tumor immunity in these individuals.
* In order to examine this issue, patients with resectable primary neoplasms involving the lungs, esophagus, or pleura will be vaccinated with autologous tumor cells exposed exvivo to decitabine and radiation following completion of appropriate combined modality therapy. Vaccine will be administered in conjunction with ISCOMATRIX adjuvant and oral celecoxib.

Primary Objective:

- To assess the safety of an epigenetically modified autologous tumor cell vaccine in conjunction with celecoxib.

Eligibility:

* Patients with histologically or cytologically proven or clinically evident primary pulmonary carcinoma or sarcoma, esophageal cancer, thymic carcinoma or malignant pleural mesothelioma undergoing resection of their neoplasms.
* Patients must be 18 years or older with an ECOG performance status of 0 2, with adequate pulmonary and cardiac function and laboratory values within normal limits.

Design:

* Patients with operable lung and esophageal carcinoma/sarcoma, thymoma, thymic carcinoma or malignant pleural mesothelioma will undergo resection of their malignancies at the NCI.
* Portions of the resected tumors will be transferred to the Thoracic Oncology Laboratory and cells will be processed to establish a cancer cell line.
* Following recovery from surgery and appropriate adjuvant chemotherapy and/or radiation, patients will be vaccinated with epigenetically-modified autologous tumor cells periodically over 6 months in conjunction with oral celecoxib.
* Systemic toxicities and delayed type hypersensitivity responses to autologous tumor cells and serologic responses to a variety of CT antigens will be assessed before and after vaccination.
* Patients will be followed with routine staging scans until disease recurrence.
* As the exact set of comparisons and analyses to be performed will be determined following completion of the trial, and will be based on limited numbers of patients, the analyses will be considered exploratory and hypothesis generating rather than definitive.
* Approximately 120 patients will be accrued to this trial in order to obtain up to 30 evaluable patients.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

INCLUSION CRITERIA PRIOR TO SURGERY (SCREENING CONSENT):

1. Patients with resectable clinically evident or histologically proven primary small cell or non-small cell lung cancers, esophageal cancers, thymoma, thymic carcinoma, primary sarcoma of the chest, or pleural mesotheliomas are eligible for treatment.
2. Patients with intracranial metastases, which have been treated by surgery or radiation therapy may be eligible for study provided there is no evidence of active disease.
3. Patients with prior Decitabine exposure are eligible for study.
4. Patients must have an ECOG performance status of 0 2.
5. Patients must be 18 years of age or older due to the unknown effects of immunologic responses to germ cell-restricted gene products during childhood and adolescent development.
6. Seronegative for HIV antibody. Note: The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus may be less responsive to the experimental treatment.
7. Seronegative for active hepatitis B, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
8. Patients must be aware of the neoplastic nature of their illnesses, the experimental nature of the therapy, alternative treatments, potential benefits, and risks.
9. Patients must be willing to sign an informed consent, and undergo resection of their malignancies at the NCI, to ensure vaccine development.

INCLUSION CRITERIA FOR TREATMENT PHASE OF PROTOCOL (STANDARD CONSENT):

1. Patients must have signed the Screening Consent
2. NCI Laboratory of Pathology confirmation of diagnosis of primary small cell or nonsmall cell lung cancers, esophageal cancers, thymoma, thymic carcinoma, primary sarcoma of the chest, or pleural mesotheliomas must have been obtained
3. Patients who were initially rendered NED by surgical resection must remain NED at the time of treatment.
4. Patients with no more than 3 intracranial metastases, which have been definitively treated by surgery or radiation therapy may be eligible for the study, provided there is no evidence of active disease for at least 2 months and no requirement for anticonvulsant therapy or steroids following treatment.
5. Patients must have an ECOG performance status of 0 2.
6. Patients must have evidence of adequate bone marrow reserve, hepatic and renal function as evidenced by the following laboratory parameters:

   * Absolute neutrophil count greater than 1500/mm(3)
   * Platelet count greater than 100,000/mm(3)
   * Hemoglobin greater than 8g/dl ( patients may receive transfusions to meet this parameter
   * PT within 2 seconds of the ULN
   * Total bilirubin <1.5 times upper limits of normal
   * Serum creatin ine less than or equal to 1.6 mg/ml or the creatinine clearance must be greater than 70 ml/min/1.73M(2).

f. Seronegative for HIV antibody. Note: The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus may be less responsive to the experimental treatment.

g. Seronegative for active hepatitis B, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.

h. Patients must be willing to practice birth control during and for four months following treatment.

i. Patients must be willing to sign the standard informed consent.

EXCLUSION CRITERIA FOR TREATMENT PHASE OF PROTOCOL:

1. Patients unable/unwilling to undergo resection of their malignancies at the NCI will be excluded.
2. Patients who are initially rendered NED by combined modality therapy but exhibit disease progression prior to initiation of vaccination will be excluded from the treatment portion of the study.
3. Patients who will have received more than two systemic cytotoxic treatment regimens for their thoracic malignancy by the time vaccination commences will be excluded.
4. Patients requiring corticosteroids (other than inhaled) will be excluded.
5. Patients with life expectancy less than 12 months will be excluded.
6. Patients receiving warfarin anticoagulation, who cannot be transferred to other agents such as enoxaparin or dabigatran, and for whom anticoagulants cannot be held for up to 24 hours will be excluded.
7. Patients with uncontrolled hypertension (>160/95), unstable coronary disease evidenced by uncontrolled arrhythmias, unstable angina, decompensated CHF (>NYHA Class II), or myocardial infarction within 6 months of study will be excluded.
8. Patients with other cardiac diseases may be excluded at the discretion of the PI following consultation with Cardiology consultants.
9. Patients with any of the following pulmonary function abnormalities will be excluded: FEV, < 30% predicted; DLCO < 30% predicted (post-bronchodilator); pO2 < 60% or pCO2 greater than or equal to 50 on room air arterial blood gas.
10. Pregnant and/or lactating women will be excluded due to the unknown, potentially harmful effects of immune response to CT-X antigens and stem cell proteins that may be expressed in placenta, fetus, and neonates.
11. Patients with active infections, including HIV, will be excluded, due to unknown effects of the vaccine on lymphoid precursors.
12. Patients with any type of primary immunodeficiencies will be excluded from the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-12-01; Primary Completion 2016-06-13 (Actual); Study Completion 2016-06-13 (Actual)

PRIMARY OUTCOMES:
Tabulation of patient toxicities and their grades | 30 days after last vaccine (up to 25 months)months)

SECONDARY OUTCOMES:
Number of patients of the first 10 sarcoma, mesothelioma and esophageal CA patients respectively with cell line development greater than or equal to 3 | When 10 patients each of the other tumor types have been recruitedother tumor types have beenrecruited
Enumeration and description of immune responses | 2 years after initial vaccination
Number of patients of first 20 lung CA patients with cell line development greater than or equal to 5. | when 20 lung cancer patients have been recruitedhave been recruited

CONTACTS AND LOCATIONS:
Overall Officials: David S Schrump, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Schrump DS, Fischette MR, Nguyen DM, Zhao M, Li X, Kunst TF, Hancox A, Hong JA, Chen GA, Pishchik V, Figg WD, Murgo AJ, Steinberg SM. Phase I study of decitabine-mediated gene expression in patients with cancers involving the lungs, esophagus, or pleura. Clin Cancer Res. 2006 Oct 1;12(19):5777-85. doi: 10.1158/1078-0432.CCR-06-0669. PMID 17020984
- [Background] Nemunaitis J, Jahan T, Ross H, Sterman D, Richards D, Fox B, Jablons D, Aimi J, Lin A, Hege K. Phase 1/2 trial of autologous tumor mixed with an allogeneic GVAX vaccine in advanced-stage non-small-cell lung cancer. Cancer Gene Ther. 2006 Jun;13(6):555-62. doi: 10.1038/sj.cgt.7700922. PMID 16410826
- [Background] Guo ZS, Hong JA, Irvine KR, Chen GA, Spiess PJ, Liu Y, Zeng G, Wunderlich JR, Nguyen DM, Restifo NP, Schrump DS. De novo induction of a cancer/testis antigen by 5-aza-2'-deoxycytidine augments adoptive immunotherapy in a murine tumor model. Cancer Res. 2006 Jan 15;66(2):1105-13. doi: 10.1158/0008-5472.CAN-05-3020. PMID 16424047